CLINICAL TRIAL: NCT04134767
Title: Kentucky Communities and Researchers Engaging to Halt the Opioid Epidemic (CARE2HOPE) - UH3 PHASE
Brief Title: Kentucky Communities and Researchers Engaging to Halt the Opioid Epidemic (CARE2HOPE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: April M Young (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Appalachian Regional Commission (Other); Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency); Centers for Disease Control and Prevention (U.S. Federal Agency); Emory University (Other)
Responsible Party: Sponsor-Investigator, April M Young, Associate Professor, Department of Epidemiology, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 52439; 4UH3DA044798-03 (NIH)
Record Dates: First submitted 2019-10-11; First posted 2019-10-22 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Substance Use; HIV Infections; HCV Infection; Sexually Transmitted Infections (Not HIV or Hepatitis); Overdose, Drug; Opioid Use
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections; Hepatitis C; Sexually Transmitted Diseases; Hepatitis; Drug Overdose

STUDY DESIGN:
Intervention Model Description: Community randomized trial. Six counties will be randomized to start 6 months of enrollment into an intervention condition. Six other communities will be assigned to 6 months of a comparison condition. All participants in both the intervention and comparison conditions will be followed for 6 months for data collection.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Linkage (Experimental): Research staff will: 1) meet with participants in person or virtually to ask questions about drug use and related behaviors, service access, and personal goals; provide overdose education and help develop a plan for reducing risks and accessing services; conduct drug testing, offer HIV and HCV testing and counseling, naloxone, and harm reduction supplies, and connection with needed services; 2) follow up with participants monthly for three months to help overcome challenges; and 3) six months post-enrollment, contact participants to conduct drug testing. Participants will complete surveys at baseline, 3 months, and 6 months
  Interventions: Behavioral: Health Linkage; Behavioral: Overdose Education
- Overdose Education (Other): The investigators will initiate the comparison group in Group 2 counties six months before the intervention begins. Research staff will conduct an overdose intervention with the comparison cohort. This will occur pre-release if individual is recruited in jail. The comparison group participants will watch a video on preventing, recognizing, and responding effectively to an opioid OD, accompanied by information about Kentucky's Good Samaritan Law and Naloxone Access Law. Research staff will answer questions after the video. Individuals will receive a Community Resource Guide at this visit.
  As in the intervention group, the comparison group participants will complete surveys at the baseline (in jail if recruited in jail, in a community setting if recruited in the community), and at 3 months and 6 months after the baseline. Surveys will be identical to those delivered to the intervention cohort.
  Interventions: Behavioral: Overdose Education

INTERVENTIONS:
Behavioral: Health Linkage — Research staff will: 1) help participants set goals and reduce their health risks by helping them to reflect on personal drug use, sexual relationships, and their consequences in the context of personal values and goals; 2) help link participants to services that they need and want; 3) offer participants the option of HIV and hepatitis C testing, provide the test result, and provide post-test counseling; and 4) provided participants nasal spray naloxone (Narcan) to carry with them in case they encounter someone who has an opioid overdose or in case they have an opioid overdose and a friend can use the naloxone to respond.
  Arms: Health Linkage
Behavioral: Overdose Education — Participants will complete a 10-minute overdose education training video on preventing, recognizing, and responding effectively to an opioid OD.

SUMMARY:
This study will test the effects of an intervention to reduce substance use and related harms among people leaving rural jails or otherwise involved in the criminal justice system. This study will compare people in a health linkage intervention with people who will get overdose (OD) education. Everyone will take part in the baseline and follow-up surveys and receive OD education. Participants will be assigned to one of the two groups by chance based on when they are enrolled to the study and if their county is randomly assigned to an intervention or a comparison condition. By doing this study, the investigators hope to learn if providing linkage to health services along with HIV, hepatitis C virus (HCV), and overdose education to people leaving rural jails or otherwise involved in the criminal justice system will reduce substance use and related harms.

DETAILED DESCRIPTION:
The overarching objective of this study is to determine the effectiveness of an evidence-based community response project using a community randomized trial. Specifically, the investigators will test the effect of an intervention to reduce substance use and related harms among people re- entering the community from rural jails or otherwise recently involved in the criminal justice system (out on bond, under warrant for arrest, arrested, on pre-trial supervision, probation or parole, court-involved, or under home incarceration with digital monitoring). This study will compare people in a health navigation intervention with a comparison group of people who will get overdose education. Everyone will take part in follow-up surveys for up to 6 months after release. The intervention is a health navigation intervention designed to reduce substance use disorder (SUD) and increase engagement in the SUD care cascade; reduce vulnerability to HIV, sexually transmitted infections (STIs), and HCV and increase engagement in the HIV, STI, and HCV care cascades; and reduce vulnerability to overdose deaths among adults who use drugs and are leaving local jails or otherwise involved in the criminal justice system. The intervention is based on enhancements to START, a Center for Disease Control-recognized, evidence-based, individual-level intervention designed to reduce HIV/STI/HCV risk.

START core components: (1) Hold pre- and post-release program sessions with clients transitioning back to the community from a correctional setting; (2) Use a client-focused incremental risk reduction approach; (3) Use assessment & documentation tools to provide structure; (4) Hire program staff that are familiar with HIV/STIs/HCV prevention and with the specific needs of people being released; (5) Staff /client relationships must be maintained post-release; (6) Conduct enrollment and schedule two pre-release program sessions within 60 days of a client's release that: a. give HIV/STI/HCV information; b. review client's HIV/STI/HCV risk; c. identify transitional needs; d. develop a personalized risk reduction and transitional plan; e. make facilitated referrals; 7) Schedule four post-release sessions to review and update the risk reduction/ transitional plan(s) and provide facilitated referrals; (8) Provide condoms at each post-release session; (9) Actively maintain contact with clients.

The investigators will modify START a priori as follows: 1) Though originally designed for young men, START has been successfully applied to women leaving correctional settings. The investigators will implement START with all genders; 2) START originally targeted incarcerated people preparing to leave correction facilities. The investigators will continue to target individuals who are incarcerated but also expand the target population to people who are involved in other parts of the criminal justice system (e.g., those out on bond, under warrant for arrest, arrested, court-involved; those on probation, parole or pre-trial supervision; and individuals under home incarceration with digital monitoring [an ankle monitoring program]). Individuals who are not incarcerated will be recruited in the communities. 3) All intervention sessions will be conducted in the community setting (post-release for those recruited in jails). 4) START's post-release sessions primarily occurred in homes and community venues, such as restaurants. Staff who will deliver START will be stationed primarily within the local department of health (DOH); 5) To enhance START's impact on drug use and HIV/HCV-related harms (e.g., drug injection frequency), the investigators will integrate the NIDA (National Institute on Drug Abuse) Standard HIV intervention into START, including rapid HIV and HCV antibody testing and counseling. In addition, START interventionists will distribute harm reduction supplies at the first intervention session with people who inject drugs (PWID). The NIDA Standard has been demonstrated to reduce drug use frequency, high-risk injection practices, and sexual risk; 6) START was not designed to reduce overdoses. The investigators will integrate an interactive training with animated scenarios and narration on preventing, recognizing, and responding effectively to an opioid OD. Participants in the intervention group will receive naloxone (not all participants will get naloxone), at their first intervention session. Interventionists will encompass OD in risk reduction motivational interviewing. 7) To accommodate participants who are not able to visit the study office in-person, data collection and intervention sessions will be conducted remotely via phone or videoconferencing.

CARE2HOPE covers the following counties: Rowan, Bath, Morgan, Menifee, Elliott, Lee, Owsley, Wolfe, Perry, Letcher, Leslie, Knott. Research staff will recruit participants from a) jails, b) Probation, Parole and Pre-Trial Services c) digital jails (i.e. home incarceration with digital monitoring programs); d) peer referral; e) existing participants in CARE2HOPE and other University of Kentucky studies, including PROUD-R2 (Peer-Based Retention of People Who Use Drugs in Rural Research) and SNAP (Social Networks among Appalachian People), who have consented to be contacted to learn about future studies; f) harm reduction and social service programs serving people who use drugs; and g) community-based organizations serving the 12 CARE2HOPE counties. Recruitment in jails will involve jails either located in CARE2HOPE counties or counties that have contracts with them to incarcerate their residents. The intervention sessions and data collection will be delivered by research staff called "Rural Health Navigators" or "REHNs". Participants are assigned to one of the two groups by chance based on when they are enrolled to the study and when their county is randomly chosen to start the project. Counties were originally randomized using a stepped wedge design. The counties were then randomized in November 2020, accounting for a new study design. The investigators randomized 12 study counties to two groups. In Months 1-6 six counties randomly assigned to Group 1 will recruit participants to the intervention, while in the remaining six counties (Group 2) the participants will be enrolled into a control condition. The investigators anticipate an average enrollment of 40 participants per county per arm, with a total final sample size for the trial of 960 (n=480intervention, n=480comparison). After a county has met its target enrollment in both conditions, the intervention and comparison activities will no longer be offered in that county.

Originally, the CARE2HOPE trial gathered data in three waves: at baseline, before the intervention had been delivered in the intervention counties; at three months post baseline, just after the intervention had been completed; and at six months post baseline, to support analyses of intervention decay. On June 24th 2022, the CARE2HOPE Data Safety Monitoring Board (DSMB) met to determine whether the trial could limit data collection to two waves - baseline and the 3-month follow up - and still ethically meet its aims. The DSMB voted to drop the six-month wave of data collection recognizing that:

1. Ending data collection at 3 months permitted the trial to test intervention effectiveness, given that the intervention itself lasted <3 months.
2. The shortened follow-up period allowed the trial to continue to enroll new participants for an additional 3 months, thus increasing capacity to generate a sufficient sample size to power analyses.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18 or older; and
* A resident of one of the 12 CARE2HOPE (C2H) counties randomized to intervention or control data collection; and
* Have used opioids to get high in the past 30 days or have injected any drug to get high during that same period (if incarcerated at home under digital monitoring program or on probation or parole: have used opioids to get high or injected any drug to get high in 30 days before the date of incarceration or start of the probation or parole term); and
* Have been recently involved in the criminal justice system defined as being incarcerated in jail or prison, out on bond, under warrant for arrest, arrested, under pre-trial supervision, on probation or parole, court-involved, or individuals who are incarcerated at home under an electronic monitoring program (i.e., digital jail) in the past 30 days.

OR

* Be a resident of or anticipate being released to one of the 12 CARE2HOPE counties randomized to intervention or control data collection; and
* Have used opioids to get high in the 30 days before they were incarcerated, or have injected any drug to get high during that period; and
* Be aged 18 or older; and
* Be incarcerated in a local jail and expected to be released in <21 days

OR

* Be a participant in the CARE2HOPE longitudinal survey who consented to be contacted for future research; and
* Be a resident of or anticipate being released to one of the 12 CARE2HOPE counties randomized to intervention or control data collection; and
* Have used opioids to get high in the 30 days before they were incarcerated, or have injected any drug to get high during that period; and
* Be aged 18 or older; and
* Be incarcerated in a local jail and expected to be released in <21 days

Exclusion criteria:

1. Previously enrolled in the START-C2H study (i.e., cannot enroll more than once)
2. Not speaking English fluently
3. Residence in or move to a county not randomized to intervention or control data collection within 21 days of release
4. Transfer to prison
5. Being charged with a violent crime (e.g., homicide, murder, rape and sexual assault, robbery, and assault)
6. Having been incarcerated for one year or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: April M Young, PhD, MPH, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from the University of Kentucky are required to be submitted to the University of Washington as part of the NIH-funded Rural Opioid Initiative (ROI) data harmonization project. The University of Washington Data Harmonization Coordinating Center (DCC) will be harmonizing data across 8 ROI studies in order to create new, harmonized datasets to be used for analyses across the consortium. The University of Washington and other ROI grantees will perform data analyses on these data for peer-reviewed publication. The harmonized datasets will be provided to other ROI grantees as required for analysis and will be considered under the umbrella of mandated DCC activities. No third parties outside of the ROI will be given access to this harmonized data. Harmonized datasets will be built to specific project concept proposals, and all project proposals must be reviewed and approved by the ROI consortium's Publications Working Group before distribution of the customized dataset.

REFERENCES:
- [Derived] Kesich Z, Ibragimov U, Komro K, Lane K, Livingston M, Young A, Cooper HLF. "I'm not going to lay back and watch somebody die": a qualitative study of how people who use drugs' naloxone experiences are shaped by rural risk environment and overdose education/naloxone distribution intervention. Harm Reduct J. 2023 Nov 10;20(1):166. doi: 10.1186/s12954-023-00900-z. PMID 37946233
- [Derived] Kesich Z, Ibragimov U, Komro K, Lane K, Livingston M, Young A, Cooper H. "I'm not going to lay back and watch somebody die": A qualitative study of how people who use drugs' naloxone experiences are shaped by rural risk environment and naloxone distribution/overdose education intervention. Res Sq [Preprint]. 2023 Sep 6:rs.3.rs-3310319. doi: 10.21203/rs.3.rs-3310319/v1. PMID 37720025

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: C2H Counties
Groups:
- Health Linkage: Research staff will: 1) meet with participants in person or virtually to ask questions about drug use and related behaviors, service access, and personal goals; provide overdose (OD) education and help develop a plan for reducing risks and accessing services; conduct drug testing, offer HIV and Hepatitis C (HCV) testing and counseling, naloxone, and harm reduction supplies, and connection with needed services; 2) follow up with participants monthly for three months to help overcome challenges; and 3) six months post-enrollment, contact participants to conduct drug testing. Participants will complete surveys at baseline, 3 months, and 6 months
  Health Linkage: Research staff will: 1) help participants set goals and reduce their health risks by helping them to reflect on personal drug use, sexual relationships, and their consequences in the context of personal values and goals; 2) help link participants to services that they need and want; 3) offer participants the option of HIV and hepatitis C testing, provide the test result, and provide post-test counseling; and 4) provided participants nasal spray naloxone (Narcan) to carry with them in case they encounter someone who has an opioid overdose or in case they have an opioid overdose and a friend can use the naloxone to respond.
  Overdose Education: Participants will complete a 10-minute overdose education training video on preventing, recognizing, and responding effectively to an opioid OD.
- Overdose Education: The investigators will initiate the comparison group in Group 2 counties six months before the intervention begins. Research staff will conduct an overdose intervention with the comparison cohort. This will occur pre-release if individual is recruited in jail. The comparison group participants will watch a video on preventing, recognizing, and responding effectively to an opioid OD, accompanied by information about Kentucky's Good Samaritan Law and Naloxone Access Law. Research staff will answer questions after the video. Individuals will receive a Community Resource Guide at this visit.
  As in the intervention group, the comparison group participants will complete surveys at the baseline (in jail if recruited in jail, in a community setting if recruited in the community), and at 3 months and 6 months after the baseline. Surveys will be identical to those delivered to the intervention cohort.
  Overdose Education: Participants will complete a 10-minute overdose education training video on preventing, recognizing, and responding effectively to an opioid OD.
Period: Overall Study
Arm/Group | Health Linkage | Overdose Education
Started | 111; 6 C2H Counties | 123; 6 C2H Counties
Completed | 67; 6 C2H Counties | 81; 6 C2H Counties
Not Completed | 44; 0 C2H Counties | 42; 0 C2H Counties
Not completed — Death | 0 | 1
Not completed — Removed for harassing staff | 0 | 1
Not completed — Lost to Follow-up | 44 | 40

BASELINE CHARACTERISTICS:
Population: One participant from the Health Linkage Arm did not have demographic data available
Units Other Than Participants: C2H Counties
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Linkage | Overdose Education | Total
Number analyzed (Participants) | 110 | 123 | 233
Number analyzed (C2H Counties) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (8.4) | 38.4 (7.1) | 37.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 63 | 121
  Male | 52 | 60 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 107 | 122 | 229
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 106 | 120 | 226
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 110 | 123 | 233

OUTCOME MEASURES:

1. Primary Outcome: Change in Substance Use Frequency
Description: Item:Self-reported frequency of substance use to get high in past 30 days (continuous variable)
  Source: Rural opioid initiative (ROI Harmonized UG3 Survey) Harmonized UG3 Survey
Time Frame: assessed at 3 months and 6 months after the baseline, change at 3 months reported
Population: The section of the baseline data instrument that captured baseline substance use was corrupted for one intervention arm participant, therefore they could not be included in the outcome assessment. During the trial, the Data Safety Monitoring Board (DSMB) approved the follow-up period to be shortened from six to three months (see Study Description for rationale).
Measure: Mean (95% Confidence Interval); unit: Days of drug use
Arm/Group | Health Linkage | Overdose Education
Number analyzed (Participants) | 66 | 81
Days of drug use | -11.2 [-14.8 to -7.7] | -5.5 [-8.4 to -2.6]

2. Secondary Outcome: Change in Engagement in HIV Risk Behaviors - Receptive Syringe Sharing
Description: Item: Self-reported recent (past 30 days) frequency of engaging in the HIV risk behavior of using a syringe that had been previously used by someone else (continuous; number and proportion)
  Source: ROI Harmonized UG3 Survey
Time Frame: assessed at 3 months and 6 months after the baseline, change at 3 months reported
Population: N = 107 injecting at baseline (those with missing N/A responses due to no injection at 3 month follow up categorized as receptive syringe sharing = 0 at follow up).
  During the trial, the DSMB approved the follow-up period to be shortened from six to three months (see Study Description for rationale).
Measure: Mean (95% Confidence Interval); unit: Receptive syringe shares
Groups:
- Health Linkage: Research staff will: 1) meet with participants in person or virtually to ask questions about drug use and related behaviors, service access, and personal goals; provide overdose education and help develop a plan for reducing risks and accessing services; conduct drug testing, offer HIV and HCV testing and counseling, naloxone, and harm reduction supplies, and connect them with needed services; 2) follow up with participants monthly for three months to help them overcome challenges; and 3) six months post-enrollment, contact participants to conduct drug testing. Participants will complete surveys at baseline, 3 months, and 6 months
  Health Linkage: Research staff will: 1) help participants set goals and reduce their health risks by helping them to reflect on personal drug use, sexual relationships, and their consequences in the context of personal values and goals; 2) help link participants to services that they need and want; 3) offer participants the option of HIV and hepatitis C testing, provide the test result, and provide post-test counseling; and 4) provided participants nasal spray naloxone (Narcan) to carry with them in case they encounter someone who has an opioid overdose or in case they have an opioid overdose and a friend can use the naloxone to respond.
  Overdose Education: Participants will complete a 10-minute overdose education training video on preventing, recognizing, and responding effectively to an opioid OD.
Arm/Group | Health Linkage | Overdose Education
Number analyzed (Participants) | 40 | 67
Receptive syringe shares | -4.0 [-9.0 to 1.0] | 5.1 [-7.0 to 17.3]

3. Secondary Outcome: Change in Engagement in HIV Risk Behaviors - Condomless Sex
Description: Item: Self-reported recent (past 30 days) frequency of condomless anal or vaginal sex (continuous; number and proportion)
  Source: ROI Harmonized UG3 Survey
Time Frame: assessed at 3 months and 6 months after the baseline, change at 3 months reported
Population: N = 133 (condomless sex item derived from baseline 2, there were n=137 participant IDs in both baseline 2 and 3-month follow up - 10 fewer than in baseline 1 and 3 month follow-up; those reporting 0 sex partners categorized as condomless sex = 0, 4 subject IDs did not report a number of sex partners and skipped condomless sex item thus n = 133) During the trial, the DSMB approved the follow-up period to be shortened from six to three months (see Study Description for rationale).
Measure: Mean (95% Confidence Interval); unit: Number of times had condomless sex
Arm/Group | Health Linkage | Overdose Education
Number analyzed (Participants) | 58 | 75
Number of times had condomless sex
  all participants | -0.7 [-3.9 to 2.5] | -1.7 [-4.6 to 1.3]
  participants with > 1 sex partner: number analyzed (Participants) | 36 | 50
  participants with > 1 sex partner | -0.4 [-4.0 to 3.2] | -2.0 [-5.9 to 1.8]

4. Secondary Outcome: Change in Engagement in HCV Risk Behaviors - Receptive Syringe Sharing
Description: Item: Self-reported recent (past 30 days) frequency of engaging in the hepatitis C risk behavior of using a syringe that had been previously used by someone else (continuous; number and proportion) Source: ROI Harmonized UG3 Survey
Time Frame: assessed at 3 months and 6 months after the baseline, change at 3 months reported
Population: N = 107 injecting at baseline (those missing N/A responses due to no injection at 3 month follow up categorized as receptive syringe sharing = 0 at follow up) During the trial, the DSMB approved the follow-up period to be shortened from six to three months (see Study Description for rationale).
Measure: Mean (95% Confidence Interval); unit: Receptive syringe shares
Arm/Group | Health Linkage | Overdose Education
Number analyzed (Participants) | 40 | 67
Receptive syringe shares | -4.0 [-9.0 to 1.0] | 5.1 [-7.0 to 17.3]

5. Secondary Outcome: Change in Engagement in HCV Risk Behaviors - Shared Injection Equipment
Description: Item: Self-reported recent (past 30 days) frequency of shared cookers, cotton, spoon, or water (continuous; number and proportion)
  Source: ROI Harmonized UG3 Survey
Time Frame: assessed at 3 months and 6 months after the baseline, change at 3 months reported
Population: N = 107 injecting at baseline (those missing N/A responses due to no injection at 3 month follow up categorized as shared injection equipment = 0 at follow up) During the trial, the DSMB approved the follow-up period to be shortened from six to three months (see Study Description for rationale).
Measure: Mean (95% Confidence Interval); unit: Number of times shared equipment
Arm/Group | Health Linkage | Overdose Education
Number analyzed (Participants) | 40 | 67
Number of times shared equipment | -10.6 [-18.2 to -3.0] | 4.5 [-7.7 to 16.8]

6. Secondary Outcome: Change in Frequency of Opioid Overdose
Description: Item:Self-reported recent (past 90 days) number of times overdosed (ordinal, continuous)
  Source: Modified from ROI Harmonized UG3 Survey
Time Frame: assessed at 3 months and 6 months after the baseline, change at 3 months reported
Population: N = 144 (those that NEVER overdosed and skipped past 90 day overdose categorized as 0 overdoses in past 90 days , n = 3 missing ever overdosed AND past 90 day overdose) During the trial, the DSMB approved the follow-up period to be shortened from six to three months (see Study Description for rationale).
Measure: Mean (95% Confidence Interval); unit: Number of times overdosed
Arm/Group | Health Linkage | Overdose Education
Number analyzed (Participants) | 64 | 80
Number of times overdosed | -0.25 [-0.6 to 0.10] | -0.59 [-1.2 to 0.02]

7. Secondary Outcome: Change in Frequency of Receptive Syringe Sharing
Description: Item:Self-reported recent (past 30 days) frequency of using a syringe that had been previously used by someone else (continuous; number and proportion)
  Source: ROI Harmonized UG3 Survey
Time Frame: assessed at 3 months and 6 months after the baseline, change at 3 months reported
Population: N = 107 injecting at baseline (those with missing N/A responses due to no injection at 3 month follow up categorized as receptive syringe sharing = 0 at follow up) During the trial, the DSMB approved the follow-up period to be shortened from six to three months (see Study Description for rationale).
Measure: Mean (95% Confidence Interval); unit: Receptive syringe shares
Arm/Group | Health Linkage | Overdose Education
Number analyzed (Participants) | 40 | 67
Receptive syringe shares | -4.0 [-9.0 to 1.0] | 5.1 [-7.0 to 17.3]

8. Secondary Outcome: Change in Frequency of Injection Drug Use
Description: Item: Self-reported recent (past 30 days) frequency of injection (ordinal, continuous)
  Source: ROI Harmonized UG3 Survey
Time Frame: assessed at 3 months and 6 months after the baseline, change at 3 months reported
Population: N = 107 injecting at baseline (those with missing N/A responses due to no injection at 3 month follow up categorized as injection times = 0 at follow up) During the trial, the DSMB approved the follow-up period to be shortened from six to three months (see Study Description for rationale).
Measure: Mean (95% Confidence Interval); unit: Number of times injected drugs
Arm/Group | Health Linkage | Overdose Education
Number analyzed (Participants) | 40 | 67
Number of times injected drugs | -33.7 [-49.2 to -18.3] | -19.5 [-30.2 to -8.7]

9. Secondary Outcome: Change in Number of Days Carrying Naloxone
Description: Item:Self-reported recent (past 90 days) number of days carrying naloxone (continuous)
  Source: Modified from ROI Harmonized UG3 Survey
Time Frame: assessed at 3 months and 6 months after the baseline, change at 3 months reported
Population: N=99 (If subject IDs had naloxone at home but missing/NA for carrying naloxone, at home response was counted to reduce missing; 46 subject IDs did NOT have a response to categorize on BOTH baseline Naloxone possession items - carrying [don't know, refuse, N/A] and having it at home [don't know, refuse, skipped] so this could not be compared to the to 3 month follow up response; 1 had no response at follow-up) DSMB approved shortened follow up period from 6 to 3 months (see Study Description).
Measure: Mean (95% Confidence Interval); unit: Number of days carrying naloxone
Arm/Group | Health Linkage | Overdose Education
Number analyzed (Participants) | 40 | 59
Number of days carrying naloxone | 4.5 [-8.5 to 17.5] | 0 [-9.7 to 9.7]

10. Secondary Outcome: Change in Evidence-based Responses to a Witnessed Overdose
Description: Item: Self-reported recent (past 90 days) engagement in evidence-based responses (i.e., called 911, gave naloxone, stayed until an ambulance or police arrived, transported person to the hospital) to a witnessed overdose by self or other bystanders (nominal)
  Source: CDC NHBS Supplemental overdose items
Time Frame: assessed at 3 months and 6 months after the baseline, change at 3 months reported
Population: N = 29 witnessed an overdose at baseline AND 3-month follow up During the trial, the DSMB approved the follow-up period to be shortened from six to three months (see Study Description for rationale).
Measure: Mean (95% Confidence Interval); unit: Evidence-based responses to overdose
Arm/Group | Health Linkage | Overdose Education
Number analyzed (Participants) | 10 | 19
Evidence-based responses to overdose | 0.1 [-0.9 to 1.1] | -0.2 [-0.6 to 0.1]

11. Secondary Outcome: Change in Number of Days on Medication for Opioid Use Disorder (MOUD) Among Participants for Whom MOUD is Indicated
Description: Item:Self-reported recent (past 90 days) frequency of being on MOUD (continuous)
  Source: Modified from ROI Harmonized UG3 Survey
Time Frame: assessed at 3 months and 6 months after the baseline, change at 3 months reported
Population: N = 35 with daily opioid use at baseline and 3-month follow up (those reporting no opioid treatment in past 90 days and NA for number of days on opioid treatment categorized as MOUD days = 0) During the trial, the DSMB approved the follow-up period to be shortened from six to three months (see Study Description for rationale).
Measure: Mean (95% Confidence Interval); unit: Days on MOUD
Arm/Group | Health Linkage | Overdose Education
Number analyzed (Participants) | 26 | 38
Days on MOUD | 23.5 [-0.4 to 47.3] | 8.2 [-7.1 to 23.6]

12. Secondary Outcome: Change in Linkage to Follow-up HCV Testing Among Those Who Test HCV Antibody Positive
Description: Item:Self-reported recent (past 90 days) access to follow-up HCV RNA testing (nominal);
  (among participants that had been told ever infected with HCV at baseline - our HCV testing item is not specific to RNA testing, ALL reporting HCV diagnosis at baseline were tested at baseline)
  Source: ROI Harmonized UG3 Survey
Time Frame: assessed at 3 months and 6 months after the baseline, change at 3 months reported
Population: N = 36 (among participants that had been told ever infected with HCV at baseline, n=13 skipped the testing item at follow-up and were excluded, ALL reporting HCV at baseline were tested at baseline) During the trial, the DSMB approved the follow-up period to be shortened from six to three months (see Study Description for rationale).
Measure: Number; unit: Percent with follow-up HCV test
Arm/Group | Health Linkage | Overdose Education
Number analyzed (Participants) | 6 | 30
Percent with follow-up HCV test | -40 | -33.3

13. Secondary Outcome: Change in Linkage to Treatment Among Those Who Test HCV RNA Positive
Description: Item: Self-reported recent (past 90 days) frequency of receiving treatment among those who test RNA positive (binary)
  Source: Modified from ROI Harmonized UG3 Survey
Time Frame: assessed at 3 months and 6 months after the baseline, change at 3 months reported
Population: N = 36 (n = 49 HCV positive AND not cleared at baseline - of those 36 responded to the follow up item on seeing a medical provider for HCV in the past 90 days) During the trial, the DSMB approved the follow-up period to be shortened from six to three months (see Study Description for rationale).
Measure: Number; unit: Percent linked to treatment
Arm/Group | Health Linkage | Overdose Education
Number analyzed (Participants) | 19 | 17
Percent linked to treatment | 0 | -5.9

14. Secondary Outcome: Change in Proportion of Syringes Obtained From Syringe Service Program Among Participants Who Inject Drugs
Description: Item: Self-reported proportion of recent (past 90 days) injections that involved a new, sterile syringe obtained from a syringe service program (continuous, proportion)
  Source: ROI Harmonized UG3 Survey
Time Frame: assessed at 3 months and 6 months after the baseline, change at 3 months reported
Population: N = 69 (no. injecting at baseline AND follow-up) During the trial, the DSMB approved the follow-up period to be shortened from six to three months (see Study Description for rationale).
Measure: Mean (95% Confidence Interval); unit: Percentage of syringes obtained at SSP
Arm/Group | Health Linkage | Overdose Education
Number analyzed (Participants) | 22 | 47
Percentage of syringes obtained at SSP | 12.4 [-10.9 to 35.7] | 0 [-11.2 to 11.2]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Health Linkage | Overdose Education
All-Cause Mortality (participants affected / at risk) | 0/111 | 1/123
Serious Adverse Events (participants affected / at risk) | 10/111 | 12/123
Other Adverse Events (participants affected / at risk) | 5/111 | 27/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Health Linkage (N=111) | Overdose Education (N=123)
Emergency Room visit or Hospitalization (General disorders) | 3 | 4
Non Fatal Overdose (General disorders) | 7 | 7
Death (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Health Linkage (N=111) | Overdose Education (N=123)
Infected with hepatitis C (Infections and infestations) | 5 | 24
Believed correctional officers could hear interview (General disorders) | 0 | 1
problems with family members, friends, or partners and infected with hepatitis C (Social circumstances) | 0 | 1
Believed correctional officers could hear interview and infected with hepatitis C (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Because of the impact of the COVID-19 pandemic, we were unable to accrue the target number of participants in either the intervention counties or the comparison counties. As a result, analyses of intervention effectiveness are underpowered. Further, data related to the follow-up HCV testing outcome should be interpreted with caution; measuring RNA-based follow-up testing for HCV is too nuanced to capture via a survey item, as it can be easily misinterpreted by participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT04134767/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT04134767/ICF_000.pdf